CLINICAL TRIAL: NCT00611338
Title: Efficacy of Group Intervention to Reduce Stress Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cheryl Gore-Felton, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SU-12192007-944
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Stress Disorders, Post-Traumatic; HIV Infections
Keywords: Complementary Therapies
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; HIV Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study investigators were blind to the condition of study participants until all intervention sessions and assessments were completed. The data were coded to mask the intervention conditions for all data analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care, Wait-List Control (Active Comparator): Participants received standard medical care, which in most clinics included informational brochures provided by physicians and clinic staff. Participants were given HIV prevention information and materials in English and Spanish and were provided referrals for services. Each individual completed assessments at immediate post intervention, 3-, 6-, and 12- months. At the end of the 12-month assessment, the wait-list control participants participated in the Trauma + HIV group arm.
  Interventions: Behavioral: HIV Skills-based Prevention
- HIV Prevention (Active Comparator): Eight, 90 minute group sessions. Three of the sessions focused on health education (e.g., medication adherence, nutrition, exercise) and five focused on HIV prevention skills (e.g., condom skills, communication, social support). Each individual completed assessments at immediate post intervention, 3-, 6-, and 12- months. At the end of the 12-month assessment, the participants in this arm were given the option to receive the 3 trauma-focused sessions from the Trauma + HIV group arm.
  Interventions: Behavioral: HIV Skills-based Prevention
- HIV Prevention plus Trauma (Active Comparator): The same format as the HIV Prevention arm with eight, 90 minute group sessions. The participants received the same five HIV prevention skills sessions along with three sessions that focused on reducing trauma-related stress (e.g., breathing training, relaxation exercises, grounding exercises, coping, trauma-related triggers). Each individual completed assessments at immediate post intervention, 3-, 6-, and 12- months.
  Interventions: Behavioral: HIV Skills-based Prevention

INTERVENTIONS:
Behavioral: HIV Skills-based Prevention

SUMMARY:
This research study will examine the usefulness of groups in reducing stress and helping individuals with HIV to stay healthy and avoid problems associated with sexually transmitted diseases. We hope to discover whether being in a group is effective in reducing stress-related symptoms and promoting healthy behaviors.

DETAILED DESCRIPTION:
This is a risk reduction intervention for adults who are living with HIV, are experiencing trauma-related stress symptoms, and are at risk for HIV transmission. By first treating trauma symptoms, the effects of a skills-building HIV risk reduction intervention for adults experiencing trauma-related symptoms such as hyperarousal, dissociation, and avoidance will be enhanced. This is based on a model the proposes trauma-related symptoms have direct effects on HIV risk behavior. Therefore, the successful treatment of trauma-related symptoms will facilitate HIV risk behavior change.

ELIGIBILITY:
Inclusion Criteria:Must be 18 years or older, must be HIV-positive, report engaging in behavior that could put them at risk for HIV transmission in the past three months, report experiencing one or more trauma-related symptoms within the past three months.

Exclusion Criteria:Exclusion criteria include the presence of gross cognitive impairment, dementia, acute psychosis, or severe physical impairment that would preclude adequate comprehension of assessment material and participation in small group intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

PRIMARY OUTCOMES:
To determine if decreasing trauma-related stress symptoms improves HIV risk reduction behavior above a standard HIV risk reduction intervention alone post -intervention 3, 6, and 12 months after the group intervention sessions. | immediate post intervention, 3 months, 6 months, and 12 months
  unprotected insertive and receptive sexual intercourse
To determine if decreasing trauma-related stress symptoms improves HIV risk reduction behavior above a standard HIV risk reduction intervention alone | immediate post intervention, 3 months, 6 months, and 12 months
  Mediation effect on trauma symptoms on HIV-related risk behavior

SECONDARY OUTCOMES:
To determine whether key variables moderate the intervention's effects. | immediate post intervention, 3 months, 6 months and 12 months
  Gender, age, ethnicity, or psychological distress (e.g. , depression, anxiety) may interact with the intervention to affect risky sexual or drug-related behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Gore-Felton Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States